CLINICAL TRIAL: NCT06433453
Title: Three Dimensional Ultrasonographic Detection of Human Ovulation and Anovulation
Brief Title: Three Dimensional Ultrasonographic Detection of Human Ovulation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Angela Baerwald, Associate Professor, University of Saskatchewan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Bio 2757
Record Dates: First submitted 2024-05-15; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Ovulation Disorder
Keywords: ovulation; 3D ultrasonography
MeSH Terms: interventions — Indomethacin; Urinalysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Indomethacin (Experimental): Oral indomethacin 50 mg three times daily for 1-7 days. The administration is terminated when signs of anovulation are observed.
  Interventions: Drug: Indomethacin 50 MG; Procedure: Transvaginal ultrasound scans; Diagnostic Test: Finger prick blood test; Diagnostic Test: Urine test

INTERVENTIONS:
Drug: Indomethacin 50 MG — The medication is commenced when a preovulatory follicle is observed. It will be administered for a minimum of one day, up to a maximum of 7 days. It will be discontinued when anovulation is observed.
Procedure: Transvaginal ultrasound scans — Ultrasound scans done intermittently before and after an ovulatory or anovulatory event
Diagnostic Test: Finger prick blood test — Capillary blood extracted from a finger prick. Blood spots are collected on a specialized card, dried and frozen before reproductive hormones are assayed from them.
  Other Names: Dried blood spots
Diagnostic Test: Urine test — Early morning urine tests to assay reproductive hormones

SUMMARY:
The research aims to compare diagnosis of ovulation and anovulation in 2D and 3D ultrasonography.

DETAILED DESCRIPTION:
Thirty healthy participants will be enrolled. When their dominant ovarian follicle has a diameter of 16 mm or more, an anti-prostaglandin medication, indomethacin 30 mg, will be administered three times daily for 1-7 days. Anti-prostaglandins are known to cause anovulation. Daily 2D and 3D ultrasound scans, and urine and finger prick blood tests for reproductive hormonal assays will be performed. The medication will be discontinued once ultrasound features of anovulation are observed. These study procedures will also be carried out on days 1, 3 and 7 after anovulation.

A second cohort of 30 participants who had 2D and 3D ultrasound scans and hormonal assays in a natural cycle in a previous study (Bio 2080; NCT05531357) will also be evaluated.

These two groups represent the anovulatory and ovulatory groups, respectively, and their 2D and 3D ultrasound features will be compared. With 2D ultrasonography as a gold standard, the study aims to determine if 3D ultrasonography improves ovulation assessment and improves the recognition of anovulatory follicles in infertility treatment

ELIGIBILITY:
Inclusion Criteria:

* Healthy biological females
* Regular menstrual cycles (21-35 days)

Exclusion Criteria:

* BMI <18 or >30
* Pregnancy
* Breastfeeding mothers
* History of infertility
* History of hysterectomy or oophorectomy
* Reproductive health issues that can interfere with study outcomes
* Smoking
* Not on any hormonal medication that affects reproduction (including hormonal contraception)
* History of metabolic syndrome or untreated thyroid disease
* Contra-indication to non-steroidal anti-inflammatory drug (NSAID) use. These include:
* Gastric ulcers or gastro-intestinal bleeding
* History of myocardial infarction or a coronary artery bypass
* Cerebrovascular disease
* Hypertension
* Chronic or acute renal failure
* Severe liver disease
* Nasal polyp syndrome

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Daily measures of follicle diameters in each ovary (mm) | 8-16 days
  Daily ultrasound scans to demonstrate the disappearance of a preovulatory follicle and replacement with a corpus luteum
Presence of corpus luteum (Y/N) | 8-16 days
  Daily ultrasound scans to demonstrate the preovulatory follicle transforming into a corpus luteum vs anovulatory follicle
Follicle stimulating hormone (FSH) level | 8-16 days
  FSH assay from dried blood spots and urine samples
Luteinizing hormone (LH) level | 8-16 days
  LH assay from dried blood spots and urine samples
Estradiol level | 8-16 days
  Estradiol assay from dried blood spots and urine samples
Progesterone level | 8-16 days
  Progesterone assay from dried blood spots and urine samples

SECONDARY OUTCOMES:
Ovulation score | 1 day
  A point system based on changes in follicle size, antrum size, follicle wall thickness, follicular vascularity, visualization of a rupture site, presence of irregular wall-antral borders, presence of internal echoes, visualization of a cumulus-oocyte complex, rise in serum LH, and rise in serum progesterone.
Endometrial thickness | 8-16 days
  Endometrial thickness and appearance to support the diagnosis of ovulation or ovulation failure.

CONTACTS AND LOCATIONS:
Overall Officials: Angela R Baerwald, PhD,MD,CCFP, Principal Investigator — University of Saskatchewan
Locations (1):
- Department of Obstetrics, Gynecology and Reproductive Sciences, University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No